CLINICAL TRIAL: NCT02096458
Title: An Open-Label Sensory Evaluation of Dexlansoprazole Delayed-Release Orally Disintegrating Tablets in Healthy Subjects : TAK-390MR(OD)_107
Brief Title: Sensory Evaluation of Dexlansoprazole Delayed-Release Orally Disintegrating Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-390MR(OD)_107; U1111-1152-9255 (Other: World Health Organization)
Record Dates: First submitted 2014-02-21; First posted 2014-03-26 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-02

CONDITIONS: Gastroesophageal Reflux Disease; Erosive Esophagitis; Heartburn
Keywords: Drug therapy
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Dexlansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexlansoprazole 30 mg (Experimental): Dexlansoprazole 30 mg delayed-release orally disintegrating tablets at Assessment 1 Day 1, Assessment 2 Day 1, and Assessment 3 Day 1.
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole delayed-release orally disintegrating tablets

SUMMARY:
The purpose of this study is to measure the in-vivo disintegration time of a single dexlansoprazole delayed-release orally disintegrating (OD) tablet.

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. An orally disintegrating (OD) form of dexlansoprazole is being tested to look at the average time that it takes for one tablet to disintegrate in the mouth of healthy volunteers. At the point at which the panelist would normally swallow the granules, they will record the time and expectorate the disintegrated tablet mass and not actually swallow the tablet or granules.

The study will enroll approximately 8 healthy volunteers. All participants will take one dexlansoprazole 30 mg OD tablet on up to three separate study days. No more than 60 mg of dexlansoprazole will be tested in any one day.

This single-centre trial will be conducted in the United States. The overall time to participate in this study is approximately 2 weeks. Participants will make up to 4 visits to the clinic, and will be contacted by telephone approximately 1 week after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. The male or female sensory panelist is between 25 and 80 years of age (inclusive), healthy volunteers for study participation, and is able to read, understand, and sign and date a written informed consent form (ICF) and any required privacy authorization before study participation.
2. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
3. The sensory panelist is qualified based on documented training and experience: All panelists will be provided by Senopsys, LLC: Panelists have been trained to detect, identify, recognize, and accurately describe different taste elements and flavor combinations and to measure oral disintegration times. Training is initially accomplished by tasting model compounds and learning to recognize and describe these accurately. These abilities are then honed and refined through additional experience in performing product testing.

Exclusion Criteria:

1. Has a history of any illness that, in the opinion of the investigator or the sensory panelist's general practitioner, might confound the results of the study or pose an additional risk in administering study drug(s) to the sensory panelist. This may include but is not limited to: a history of relevant drug or food allergies; history of cardiovascular or central nervous system disease; history or presence of clinically significant pathology; recent history of disease involving head, neck, esophagus (especially malignancy, radiation therapy, fungal infection where taste perception can be altered) or history of mental disease.
2. If female, the sensory panelist is pregnant, nursing, planning to become pregnant during the study.
3. Has a known hypersensitivity to dexlansoprazole or any component of dexlansoprazole delayed-release orally disintegrating (OD) tablet or proton pump inhibitor (PPI) (including lansoprazole, omeprazole, rabeprazole, pantoprazole, or esomeprazole).
4. Is currently taking any contraindicated medications.

   -

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- Woburn, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 8 participants were screened for the study, and all participants subsequently enrolled.
Groups:
- Dexlansoprazole: Single oral dose of 30 mg dexlansoprazole delayed-release orally disintegrating tablet
Period: Overall Study
Arm/Group | Dexlansoprazole
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The population consisted of all enrolled participants.
Arm/Group | Dexlansoprazole
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: Years] | 56.5 [35 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to In-Vivo Disintegration of Dexlansoprazole 30 mg Orally Disintegrating Tablets
Description: The disintegration time is the total time from when the participant places the tablet on their tongue until the time at which the participant would normally swallow the remaining materials from the disintegrated tablet. The average disintegration time will be calculated for each participant based on 3 separate tests.
Time Frame: Day 1
Population: The populations consisted of all enrolled participants.
Measure: Mean (Full Range); unit: Seconds
Arm/Group | Dexlansoprazole
Number analyzed (Participants) | 8
Seconds | 36.0 [30.7 to 39.3]

ADVERSE EVENTS:
Time Frame: Up to Day 10
Arm/Group | Dexlansoprazole
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Research Organization shall not publish any articles or papers nor make any presentations, nor assist any other person in publishing any articles or papers or in making any presentations relating or referring to the Study or any results, data or insights from or any data, information or materials obtained or generated in the performance of its obligations without the prior written consent of Takeda, which consent may be granted or withheld in Takeda's sole discretion.